CLINICAL TRIAL: NCT03496415
Title: The Neuroprotective Effect of Remote Ischemic Conditioning in Aneurysm Coiling
Brief Title: The Neuroprotective Effect of Remote Ischemic Conditioning in Aneurysm Coiling Therapy
Acronym: NEAT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, MD, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-NEAT
Record Dates: First submitted 2018-03-22; First posted 2018-04-12 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic conditioning (Experimental)
  Interventions: Device: remote ischemic conditioning
- Sham remote ischemic conditioning (Sham Comparator)
  Interventions: Device: sham remote ischemic conditioning

INTERVENTIONS:
Device: remote ischemic conditioning — Remote ischemic conditioning is performed by using an electric autocontrol device with cuffs that inflated to a pressure of 200 mm Hg during the ischemic period (Patent No. CN200820123637.X, China)
  Arms: Remote ischemic conditioning
Device: sham remote ischemic conditioning — sham remote ischemic conditioning is performed by using an electric autocontrol device with cuffs that inflated to a pressure of 60 mm Hg
  Arms: Sham remote ischemic conditioning

SUMMARY:
The overall incidence of DWI positive for thromboembolic events following endovascular treatment of intracranial aneurysms is proximately 50%. Whether remote ischemic conditioning was safe and effective to reduce ischemic brain lesions on DWI after endovascular treatment of intracranial aneurysms is still unclear. The investigators' hypothesis is that remote ischemic conditioning is a safe and effective strategy to reduce new ischemic lesions in intracranial aneurysms patients undergoing endovascular treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Unruptured brain aneurysm deemed suitable for neuroendovascular repair
* Normal baseline brain MRI
* Female subjects of childbearing potential have a negative pregnancy test.
* Signed informed consent prior to entering study

Exclusion Criteria:

* Dissecting or mycotic brain aneurysm.
* Planned endovascular vessel sacrifice as the primary modality for aneurysm treatment
* Severe, sustained hypertension (SBP > 185 mmHg or DBP > 110 mmHg)
* Contraindication for remote ischemic conditioning: severe soft tissue injury, fracture, or peripheral vascular disease in the upper limbs
* Pre-morbid modified Rankin scale score of greater than 1
* Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations
* Patients who are unable to have an MRI scan for any reason.
* Currently participating or previously participated in any investigational drug or device study within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
The presence of ≥1 new brain lesions on DWI | within 72 hours after endovascular treatment
  Assessed by DWI

SECONDARY OUTCOMES:
Number of new ischemic lesions | within 72 hours after endovascular treatment
Volume of new ischemic lesions | within 72 hours after endovascular treatment
National Institutes of Health Stroke Scale | 7 days or discharge
  Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating more severe neurologic deficits.
Cerebrovascular events | 30 days
  Cerebrovascular events included ischemic stroke, hemorrhagic stroke, and TIA.
Nondisabling events | 30 days
  Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating more severe neurologic deficits.National Institutes of Health Stroke Scale ≤3 or TIA is defined as nondisabling events
Modified Rankin Scale | 30 days
  Scores on the modified Rankin scale of functional disability range from 0 (no symptoms) to 6 (death).

OTHER OUTCOMES:
Occurrence of adverse events and serious adverse events | 30 days
  Occurrence of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Suzhou Municipal Hoapital, Suzhou, Anhui
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan
  - Shengli Oilfield Center Hospital, Dongying, Shandong
  - Nanyang City Center Hospital, Nanyang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou